CLINICAL TRIAL: NCT03436836
Title: Nalbuphine as an Adjuvant to Local Anaesthetic Mixture in Peribulbar Cataract Surgery a Randomized Controlled Study
Brief Title: Nalbuphine as an Adjuvant to Local Anaesthetic Mixture in Peribulbar Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Nadia Yossif Helmy (Unknown); Ahmed Elbadawy Mahmoud (Unknown); Abdelhamid, Bassant Mohamed, M.D. (Individual); Atef Kamel Salama (Unknown); Mostafa Abdalwahab Elberry (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia&I.C.U and Pain Clinic, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-93-2017
Record Dates: First submitted 2017-12-30; First posted 2018-02-19 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Nalbuphine as an Adjuvant to L. A in Peribulbar Block for Cataract Surgery
MeSH Terms: interventions — Nalbuphine; Lidocaine; Bupivacaine; Hyaluronoglucosaminidase; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Forty-four patients were enrolled in the current study and randomly allocated into two equal groups [Group N (n=22) and Group C (n=22)]. Two patients in Group N and three patients in Group C were excluded from the study due to failure of the block to achieve satisfactory surgical condition (inadequate akinesia OMS>2) so, received additional supplementations 2-3 ml of LA mixture and were excluded from the study
Who Masked: Participant, Care Provider
Masking Description: The enrolled patients were randomized according to computer-generated random number into two equal groups of twenty two patients each and concealed using sequentially numbered sealed opaque envelopes.
  Patients of Group N received local anesthetics received 6 ml of 0.5% bupivacaine 1 ml hyaluronidase (75 IU) , and 4mg of Nalbuphine in 1 ml of saline (total 8 ml) and patients of Group C received 6 ml of 0.5% bupivacaine, 1 ml hyaluronidase (75 IU) and1 ml saline (total 8 ml)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (Experimental): group N was received a mixture of 3 ml of 2% lidocaine, 4 ml of 0.5% bupivacaine with hyaluronidase (75IU) and 4mg of nalbuphine in 1 ml normal saline.
  Nalbuphine (20mg amp.) was prepared in 0.9% sodium chloride in 5mL syringe. If the block was inadequate after 10 minutes, a 2-4 ml supplementation of local anesthetics was given by the same technique and the patient was excluded from the study
  Interventions: Drug: Nalbuphine; Drug: lidocaine, bupivacaine , hyaluronidase
- Group C (Active Comparator): Patients of group C was received a mixture of 3 ml of 2% lidocaine, 4 ml of 0.5% bupivacaine with hyaluronidase (75 IU) and 1 ml normal saline
  Interventions: Drug: lidocaine, bupivacaine, hyaluronidase , saline

INTERVENTIONS:
Drug: Nalbuphine — Both groups received 8 ml solution for the peribulbar block, Patients of group N was received a mixture of 3 ml of 2% lidocaine, 4 ml of 0.5% bupivacaine with hyaluronidase (75IU)(16) and 4mg of nalbuphine in 1 ml normal saline. Patients of group C was received a mixture of 3 ml of 2% lidocaine, 4 ml of 0.5% bupivacaine with hyaluronidase (75 IU) and 1 ml normal saline. Nalbuphine (20mg amp.) was prepared in 0.9% sodium chloride in 5mL syringe.
  If the block was inadequate after 10 minutes, a 2-4 ml supplementation of local anesthetics was given by the same technique and the patient was excluded from the study.
  After adequate analgesia (loss of sensation to touch by a small cotton wool) and akinesia, the surgeon was allowed to start the surgery
  Arms: Group N
Drug: lidocaine, bupivacaine, hyaluronidase , saline — lidocaine, 0.5% bupivacaine, 1 ml hyaluronidase (75 IU) and 1 ml saline (total 8 ml).
  Arms: Group C
Drug: lidocaine, bupivacaine , hyaluronidase — 2% lidocaine, 4 ml of 0.5% bupivacaine with hyaluronidase (75IU)
  Arms: Group N

SUMMARY:
Nalbuphine has been used as an adjuvant to bupivacaine in intrathecal, epidural, caudal anesthesia and peripheral nerve blocks showing an increase in the efficacy and the duration of postoperative analgesia.The aim of this study is evaluation of the effect of nalbuphine when used as an adjuvant to a local anesthetic mixture in peribulbar block undergoing cataract surgery

DETAILED DESCRIPTION:
44 patients (22 in each group) scheduled for elective cataract surgery using peribulbar block. Patients of Group N received local anesthetics received 6 ml of 0.5% bupivacaine 1 ml hyaluronidase (75 IU), and 4mg of Nalbuphine in 1 ml of saline (total 8 ml) and patients of Group C received 6 ml of 0.5% bupivacaine, 1 ml hyaluronidase (75 IU) and1 ml saline (total 8 ml).

Addition of nalbuphine to bupivacaine in peribulbar block is associated with reduced the time of onset of globe akinesia, increased the duration of globe akinesia and analgesia with better postoperative pain relief

ELIGIBILITY:
Inclusion Criteria:

* patients aged 40-60 years.
* both sex.
* ASA physical status Ι&II.
* Patient with axial globe length below 26

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Coagulation abnormalities(INR>1.4).
* More than ASA II.
* High myopia with axial length more than 26 mm.
* Mentally retarded patients and failure of proper communication as in deafness .
* Morbidly obese patients(BMI>35)
* Patients with glaucoma (increased IOP>20mmgh)
* Patients with history of hypersensitivity to study drugs

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Sensory block | 12 hours Postoperative
  Duration of the sensory block

SECONDARY OUTCOMES:
Motor block | 12 hours Postoperative
  Duration of the motor block
Sensory block onset | 12 hours Postoperative
  Onset of the sensory block
Mean Arterial blood pressure | 24 hours postoperatively
  Hemodynamic parameter as mean blood pressure(mmHg)
Adverse effects of the used drugs | 24 hours postoperatively
  Adverse effects of the used drugs as nausea and vomiting
Satisfaction assessed at the end of surgical procedure by using a three-point scale | 6 hours Postoperative
  Patient satisfaction and surgeon satisfaction

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ahmed Abdalla Mohamed, Cairo
  - Ahmed Abdalla, Cairo

IPD SHARING:
Plan to Share IPD: No
Via scholar Gate